CLINICAL TRIAL: NCT03288649
Title: Qualitative Evaluation of Therapeutic Alliance in Adolescent Psychiatry: Crossing Perspectives of Adolescents, Parents and Physicians
Brief Title: Qualitative Evaluation of Therapeutic Alliance in Adolescent Psychiatry
Acronym: EVAADO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Victor Dupouy (Other)
Responsible Party: Principal Investigator, Anne Revah-Levy, Pr Anne Revah-Levy, Centre Hospitalier Victor Dupouy
Other Study IDs: 20140600001072
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Anorexia Nervosa; Depression; School Phobia
MeSH Terms: conditions — Anorexia Nervosa; Depression; Phobia, School

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorexia nervosa: adolescents with anorexia nervosa (N=20 ?), their parents (N=20), their physicians (N=20)
- Anxiety based school refusal: adolescents with anxiety based school refusal (N=20 ?), their parents (N=20), their physicians (N=20)
- Depression: adolescents with depression (N=20 ?), their parents (N=20), their physicians (N=20)

SUMMARY:
Context: Psychiatric disorders (anorexia nervosa, depression, anxiety based school refusal) are a major public health concern in adolescence. Their treatment is a challenge for the families, the health care system and society. The treatment is complex and non-standardized. In clinical practice, the relational dimension between the stakeholders is recognized by all. Nevertheless no study has ever crossed their perspectives about therapeutic alliance in adolescent psychiatry.

Objective: to explore, within a qualitative approach, how a therapeutic alliance is established in three different clinical situations according to the adolescents, their parents and their physicians by crossing their perspectives.

Methods: This is a national (France) multi-center qualitative study based on 180 semi-structured interviews. Participants (purposively selected until data saturation) came from three different sub-samples: (i) adolescents with anorexia nervosa (N =20) plus their parents (N=20) and their physicians (N=20), (ii) adolescents with depressions (N=20) plus their parents (N=20) and their physicians (N=20), and (iii) adolescents with anxiety-based school refusal (N=20) plus their parents (N=20) and their physicians (N=20). Data are collected through open ended semi structured interviews and independently analyzed with NVivo V.11 software by three researchers according to the principles of Interpretative Phenomenological Analysis.

ELIGIBILITY:
Inclusion Criteria:

* adolescents, boys and girls, aged 12 to 18 years, speaking fluent French, with (i) anorexia nervosa according to DSM 5 criteria (ii) depressive disorders (dysthymia, depressive episode) according to DSM 5 criteria (iii) anxiety-based school refusal according to four criteria:

  1. refusal to attend school (to operationalize this first criterion, adolescents were included if they had not attended school at all for at least one month before starting treatment); (2) presence of a DSM-5 anxiety disorder (except obsessive-compulsive or post-traumatic stress disorders) with emotional upset at the prospect of attending school; (3) absence of a DSM-5 conduct disorder; and (4) parental knowledge of the adolescent's whereabouts during the period of non-attendance.

     that led to treatment that had begun at least six months earlier and clinically determined to be well enough to participate in a research interview.
* receiving treatment for at least 6 months
* one parent at least agrees to participate

Exclusion Criteria:

* acute symptoms and serious somatic and/or psychiatric co-morbidities

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: adolescents with psychiatric disorders
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
to describe the facilitators of therapeutic alliance within adolescent psychiatry using a qualitative approach | 2 years
  qualitative methodology using verbal data analysis of semi-structured interviex

CONTACTS AND LOCATIONS:
Overall Officials: Anne Revah-Levy, MD PhD, Principal Investigator — Paris diderot University
Locations (2):
- France (2):
  - CHVictorDupouy, Argenteuil
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No